CLINICAL TRIAL: NCT02277964
Title: An Observational Study to Evaluate Disease Control, Safety and Immunological Changes in Patients With Relapsing Remitting Multiple Sclerosis (RRMS) Transferred From Previous Treatment With Natalizumab to Fingolimod.
Brief Title: Disease Control in RRMS Transferring Treatment From Natalizumab to Fingolimod
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: CFTY720D2324
Record Dates: First submitted 2014-10-27; First posted 2014-10-29 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: RRMS; Natalizumab; Fingolimod; Treatment Change; Disease Activity
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * assess alterations of the composition of myeloid cells and lymphocyte subpopulations (i.e. naïve, central memory and effector memory and regulatory T cells, B cells) and adhesion molecule expression in peripheral blood
  * measure autoantigen specific T cell proliferation and IFNγ production
  * characterize transcriptomic alterations (including mRNA and small non-coding RNA expression) in lymphocytes of MS-patients
  * assess changes in plasma cytokine, chemokine, and Matrix metallo-proteinase levels
  * assess the migratory capacity of PBMCs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RRMS with treatment change: All patients with treatment change from natalizumab 300mg iv monthly to fingolimod 0.5mg orally/daily.
  16 patients were switched with an interval of 8 weeks until october 2013. After an interims analysis the interval has been changed to 4 weeks (after october 2013).

SUMMARY:
This is an observational study to develop new hypothesis regarding the dynamic and safety of switching from natalizumab to fingolimod:

* Comparison of disease activity (clinical and MRI) during the year after change of therapy in comparison to the year before change
* Dynamic of onset of disease activity after having stopped treatment with natalizumab
* Change of immunological parameters during treatment change from natalizumab to fingolimod in comparison to clinical and MRI measures

DETAILED DESCRIPTION:
The risk of progressive multifocal leukoencephalopathy (PML) upon treatment with natalizumab increases over time, at least into the 3rd year of therapy. Many Multiple Sclerosis (MS) patients who are currently being treated with natalizumab, as well as their physicians, are looking for alternative MS treatments, fingolimod being one. In transferring patients from natalizumab to fingolimod, it is not known if their co-administration leads to an increased risk of adverse effects due to a shared feature that both have immunomodulation as a mechanism of action. Therefore a sufficient washout period after natalizumab discontinuation and fingolimod initiation is desirable. However, this has to be balanced with the increasing risk over time of recurring disease activity while patients are untreated.

This study prospectively evaluates how safe it is to switch patients from natalizumab to fingolimod treatment following cessation of natalizumab treatment, in a cohort of RRMS patients.

Safety of the proposed transition paradigms is defined as both traditional safety measures but also recurrence of disease activity during a washout period of 8 weeks after the cessation of natalizumab treatment followed by fingolimod treatment initiation. An interim analysis of the first 15 patients revealed a clinical and MRI activity in 38.5 and 64.3% respectively. Therefore a shorter interval was defined for any subject entering into this study after october 2013: the interval was defined to be 4 weeks for those patients.

Overall, the study aims to provide guidance to physicians on the management of natalizumab-treated patients for whom a transition to fingolimod treatment is considered an appropriate treatment alternative.

An evidence based rationale for changing to a 4 or 8 week wash out period is not possible due to missing evidence. Due to the known risk of PML for patients being treated with natalizumab for more than 2 years, starting fingolimod during natalizumab therapy seems to be inappropriate, as an elevated risk for JC Virus (JCV) manifestation could be expected in this constellation. On the other hand considerable shortening of the 8-weeks interval could be favorable to prevent clinical and MRI activity. An interval of 4 weeks between last dose of natalizumab and first dose of fingolimod seemed to be an appropriate compromise to balance risks and benefits of this treatment transition.

Fingolimod and Natalizumab are influencing the immune system in completely different ways. It is therefore highly interesting not only to monitor clinical disease activity and MRI activity, but also to study immunological responses during the switching phase of both drugs.

The change of therapy from natalizumab to fingolimod poses possible risks. On the one hand MS could reactivate if the start of fingolimod is delayed too long, on the other hand infectious problems could emerge if fingolimod is started early and the patient is treated with two concomitant immunomodulators. Analyzing the immune response during the critical Switch period may help to identify markers that predict recrudescence of disease activity or a severe suppression of the immune response. It is known that natalizumab can block migration of lymphocytes via endothelial cells by interaction with integrins. More recently, it has been described that natalizumab influences also gene expression profiles in lymphocytes and that the blockade of migration over endothelial cells might not be as constant as the clinical effect predicts.

In contrast to natalizumab, fingolimod blocks egress of lymphocytes from secondary lymphoid organs (SLO) such as lymph nodes. This effect is mediated by functional antagonization sphingosine-1-phosphate (S1P) receptors on lymphocytes by fingolimod. Due to a different expression of lymph node homing receptors naïve and central memory T-cells regularly circulate to SLO and are consequently more prone to sequestration to SLO than effector memory cells that do not circulate to SLO on a regular basis. This is reflected by a decrease of naïve and central memory cells and a relative increase of effector memory cells in peripheral blood of fingolimod treated patients. So far, the effect of a concomitant treatment of natalizumab and fingolimod on the immune system has not been studied.

The different aspects of immune modulation of both drugs will be studied. At baseline and then at early follow-up visit (8, 12, 16, 20 weeks) we aim to:

* assess alterations of the composition of myeloid cells and lymphocyte subpopulations (i.e. naïve, central memory and effector memory and regulatory T cells, B cells) and adhesion molecule expression in peripheral blood
* measure autoantigen specific T cell proliferation and Interferon gamma (IFNγ) production
* characterize transcriptomics alterations (including messenger ribonucleic acid (mRNA) and small non-coding RNA expression) in lymphocytes of MS-patients
* assess changes in plasma cytokine, chemokine, and Matrix metalloproteinase levels
* assess the migratory capacity of peripheral blood mononuclear cells (PBMCs)

For the patients being recruited after october 2013 with a shorter wash out period, the neuroimmunological analysis has been omitted.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18-65 years
* Subjects with RRMS, defined by 2010 revised McDonald criteria
* Patients with Expanded Disability Status Scale (EDSS) score of 0-6.0 inclusive
* Patients on treatment with natalizumab for at least 6 months prior to screening

Exclusion Criteria:

* Patients with serious cardiovascular conditions and/or history or presence of a second- and third-degree aortic valve (AV) block, corrected QT interval (QTc) >450 ms in males and >470 ms in females
* Patients receiving class Ia or III antiarrhythmic drugs
* Patients with proven history of sick sinus Syndrome (SSS) or sinoatrial (SA) heart block
* Patients with uncontrolled hypertension
* Patients with resting heart rate (HR) <45 bpm
* Patients who have been treated with Fingolimod or cladribine at any time
* Patients with a history of malignancy of any organ system
* Patients with severe respiratory or hepatic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with relapsing remitting multiple sclerosis, who are planned to change treatment from natalizumab to fingolimod
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2012-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Relapse rate | up to 108 Weeks
New or newly enlarging lesions/Gadolinium enhancing lesions | up to 108 Weeks

SECONDARY OUTCOMES:
Immunological markers | Weeks 0, 8, 12, 16, 20

CONTACTS AND LOCATIONS:
Overall Officials: Ludwig Kappos, Prof., MD, Principal Investigator — Department of Neurology, University Hospital Basel, Petersgraben 4, 4031 Basel, Switzerland
Locations (1):
- University Hospital Basel, Switzerland, Basel, Switzerland